CLINICAL TRIAL: NCT01119599
Title: Phase 1 Trial of RO4929097 in Combination With Standard Radiotherapy and Temozolomide for Newly Diagnosed Malignant Glioma: A Pharmacokinetic and Pharmacodynamic Study
Brief Title: RO4929097, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01410; NCI-2011-01410 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000672641; 09-177 (Other: Memorial Sloan-Kettering Cancer Center); 8556 (Other: CTEP); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-06

CONDITIONS: Acoustic Schwannoma; Adult Anaplastic (Malignant) Meningioma; Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Brain Stem Glioma; Adult Choroid Plexus Neoplasm; Adult Craniopharyngioma; Adult Diffuse Astrocytoma; Adult Ependymoblastoma; Adult Ependymoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Grade I Meningioma; Adult Grade II Meningioma; Adult Medulloblastoma; Adult Mixed Glioma; Adult Myxopapillary Ependymoma; Adult Oligodendroglioma; Adult Papillary Meningioma; Adult Pilocytic Astrocytoma; Adult Pineal Gland Astrocytoma; Adult Pineoblastoma; Adult Pineocytoma; Adult Primary Melanocytic Lesion of Meninges; Adult Subependymal Giant Cell Astrocytoma; Adult Subependymoma; Adult Supratentorial Primitive Neuroectodermal Tumor; Malignant Adult Intracranial Hemangiopericytoma
MeSH Terms: conditions — Neuroma, Acoustic; Meningioma; Astrocytoma; Ependymoma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Medulloblastoma; Glioma; Oligodendroglioma; Pinealoma; Glioma, Subependymal | interventions — Radiotherapy, Conformal; 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Radiotherapy, Intensity-Modulated; Temozolomide

ARMS (1):
- Treatment (RO4929097, surgery, radiation therapy) (Experimental): See Detailed Description.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Gamma-Secretase Inhibitor RO4929097; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temozolomide; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3-D conformal radiation therapy
  Other Names: 3-dimensional radiation therapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: RO4929097
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temodal; Temodar
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase I trial studies the side effects and best dose of gamma-secretase/Notch signalling pathway inhibitor RO4929097 (RO4929097) when given together with temozolomide and radiation therapy in treating patients with newly diagnosed malignant glioma. Enzyme inhibitors, such as gamma-secretase/Notch signalling pathway inhibitor RO4929097, may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving gamma-secretase/Notch signalling pathway inhibitor RO4929097 together with temozolomide and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose/recommended phase II dose of RO4929097 in combination with temozolomide and radiotherapy in patients with glioblastoma or malignant gliomas.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of RO4929097 when given in combination with temozolomide (correlative study C1).

II. To evaluate brain and tumor penetration of RO4929097 when given in recommended phase II single agent schedule and when given at the maximum tolerated dose (MTD) for the combination with radiotherapy and temozolomide (correlative study C2).

TERTIARY OBJECTIVES:

I. To evaluate pharmacodynamic effects of RO4929097 in the resected specimens, and comparison with specimens obtained from untreated patients.

II. Effects of RO4929097 on the cancer stem cell population (correlative study C4).

III. Effects of RO4929097 on angiogenesis (correlative study C5). IV. To evaluate the combined effects of RO4929097, radiation and temozolomide in explants established from patients' tumor specimens (correlative study C6).

V. To evaluate the effects of RO4929097 on magnetic resonance imaging (MRI) parameters (correlative study C7), including dynamic contrast enhanced (DCE) MRI perfusion, diffusion weighted imaging and volumetric analysis.

VI. Preliminary evaluation of efficacy of this treatment regimen: 6 month (6m) and median progression-free and overall survival, and response rates.

VII. To evaluate potential biomarkers of gamma-secretase and Notch inhibition activity (correlative study C8).

OUTLINE: This is a dose-escalation study of gamma-secretase/Notch signalling pathway inhibitor RO4929097. Patients are assigned to 1 of 2 treatment arms.

PRE-SURGERY TREATMENT: Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 orally (PO) once daily (QD) on days 1-7 of week 1 and day 1 of week 2.

SURGERY: Patients undergo surgery 2-3 hours after administration of gamma-secretase/Notch signalling pathway inhibitor RO4929097 on day 1 of week 2.

TREATMENT CONCURRENT WITH RADIOTHERAPY: Beginning 3-4 weeks after surgery, patients undergo conventional focal (intensity-modulated radiation therapy [IMRT] or 3-D conformal) radiotherapy 5 days a week for approximately 6 weeks. Patients also receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD for approximately 10 weeks beginning the day of radiotherapy and temozolomide PO QD for approximately 6 weeks beginning the day before radiotherapy.

ADJUVANT TREATMENT FOLLOWING RADIOTHERAPY: Approximately 4 weeks after completion of radiotherapy, patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days 1-28 and temozolomide PO QD on days 1-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed glioblastoma, anaplastic astrocytoma, gliosarcoma or other malignant gliomas with the exception of pure anaplastic oligodendroglioma; note: patients with presumed malignant glioma based on radiographic assessment may be enrolled onto Arm A of the study without histological confirmation provided they meet the following additional eligibility criteria:

  * The MRI of the brain shows typical findings of a malignant glioma or glioblastoma (single ring-enhancing mass with necrotic portions)
  * To exclude brain abscess, diffusion-weighted MRI must show absence of restricted diffusion corresponding to the necrotic center of the lesion
  * To confirm the diagnosis of neoplastic disease, MR perfusion must show that the lesion has increased perfusion
  * To exclude pilocytic astrocytoma, the patient's age must be over 25
  * To exclude brain metastasis, a computed tomography (CT) of the chest, abdomen and pelvis must demonstrate absence of other malignancy
  * The principal investigator must review MRI and CT findings and agree with diagnosis of presumed malignant glioma

    * Note: If after the on-protocol surgery the patient is found not to meet histological criteria described (diagnosis of glioblastoma, anaplastic astrocytoma, gliosarcoma or other malignant gliomas with the exception of pure anaplastic oligodendroglioma), the patient will be removed from the study and replaced
* ARM A ONLY: Patients must have an indication for additional debulking surgery as part of their initial treatment
* Life expectancy of greater than 2 months
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%)
* Hemoglobin >= 9 g/dL
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Total bilirubin < 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of RO4929097; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097
* Female patients of childbearing potential are defined as follows:

  * Patients with regular menses
  * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
  * Women who have had tubal ligation
* Female patients may be considered to NOT be of childbearing potential for the following reasons:

  * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
  * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
  * Pre-pubertal females; the parent or guardian of young female patients who have not yet started menstruation should verify that menstruation has not begun. If a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior chemotherapy, radiotherapy, biological or experimental therapy for glioma
* Prior history of radiotherapy to the brain, head or neck
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or other agents used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* Preclinical studies indicate that RO4929097 is a substrate of CYP3A4 and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Patients with known history of hepatitis B or C, or who have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible; (hepatitis B and C serology should be obtained as part of pre-treatment evaluation but are not required for eligibility)
* Patients with uncontrolled electrolyte abnormalities including hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, and hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, history of torsades de pointes or other significant cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with RO4929097 or temozolomide; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* A corrected QT (QTc) > 450 msec in males and a QTc > 470 msec in females
* Patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to prior therapy are not eligible to participate in this study
* ARM A ONLY: Patients with contraindication to a brain surgical procedure
* A requirement for antiarrhythmics or other medications known to prolong QTc

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose defined as the highest dose studied for which the incidence of dose limiting toxicity is less than 33% using National Cancer Institute Common Toxicity Criteria | 28 days
  The percentage of patients who experience toxicity at each dose level will be calculated, with a 95% confidence interval.

SECONDARY OUTCOMES:
Changes in MRI parameters | Baseline to up to 4 years
  Perfusion and diffusion-based MRI parameters including but not restricted to blood volume, mean and median apparent diffusion coefficient and structural volumes will be analyzed. Results will be summarized, and mean and median values at different time points will be tabulated. Changes in such parameters will be checked for statistical significance and correlated with the disease status.
Percent changes in serum YKL-40 levels and hair follicle HES1 levels | Baseline to up to 4 years
  Means and medians of all patients together will be calculated and tabulated for each time point, with depiction of standard deviations. A Wilcoxon test will be used to determine p value of changes in mean values of YKL-40 and hairy and enhancer of split 1, (Drosophila) (HES1), with a p value of less than 0.05 considered statistically significant.
Pharmacokinetic (PK) parameters of gamma-secretase/Notch signalling pathway inhibitor RO4929097 | Pre-dose, 30 minutes, 1, 2, 4, 6, and 8 hours
  Noncompartmental and/or compartmental methods will be used to calculate PK parameters of gamma-secretase/Notch signalling pathway inhibitor RO4929097 and temozolomide from the plasma concentration-time data collected from each individual. Descriptive statistics (including number, mean and/or median, standard deviation, coefficient of variation, and range) for PK parameters will be tabulated by dose level.

OTHER OUTCOMES:
Expression of a variety of proteins through immunohistochemistry and/or real time quantitative polymerase chain reaction and tumor tissue culture | Up to 4 years
  Analyses will include comparison of results before and after exposure to gamma-secretase/Notch signalling pathway inhibitor RO4929097 (Wilcoxon rank sum test), as well as status of the Notch pathway and cancer stem cells in a control population of 20 untreated patients (Mann Whitney test).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Omuro, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Virginia Cancer Center, Charlottesville, Virginia